CLINICAL TRIAL: NCT04152304
Title: Feasibility of the SINEX Program for Patients With Traumatic Anterior Shoulder Instability
Brief Title: Feasibility of the Sinex Program for Shoulder Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Norway University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Liv Heide Magnussen, Professor, Western Norway University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1189/REK vest
Record Dates: First submitted 2019-10-28; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Anterior Shoulder Dislocation
Keywords: shoulder instability; feasibility studies; neuromuscular exercise

STUDY DESIGN:
Intervention Model Description: Feasibility study. One group before and after design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility of the SINEX for treatment of shoulder instability (Experimental): Feasibility of the SINEX program for treatment and evaluation of of traumatic anterior shoulder instability eligible for surgery
  Interventions: Other: Sinex program (neuromuscular training program)

INTERVENTIONS:
Other: Sinex program (neuromuscular training program) — The SINEX program is a three months neuromuscular training program aiming to increase neuromuscular stability of the shoulder

SUMMARY:
An optimal treatment for traumatic anterior shoulder instability (TASI) remains to be identified. A shoulder instability neuromuscular exercise (SINEX) program has been designed for patients with TASI, but has not yet been tested in patients eligible for surgery. The purpose of this study was to investigate and evaluate the feasibility and safety of the SINEX program for patients diagnosed with TASI and eligible for surgery.

A feasibility study with an experimental, longitudinal design using both quantitative and qualitative research methods. Participants undergo the SINEX program, a twelve week exercise program including physiotherapist supervised sessions. Feasibility data on recruitment, retention, compliance, acceptability and safety was collected through observation and individual semi-structured interviews. Clinical tests and self-report questionnaires were completed at baseline and 12 weeks follow-up. Clinical assessments included apprehension and relocation tests, shoulder joint position sense (SJPS), shoulder sensorimotor control measured by center of pressure path length (COPL) on a force platform, isometric strength measured by Constant Score - Isometric Maximal Voluntary Contraction (CS-iMVC), self-report questionnaires included Western Ontario Shoulder Instability Index (WOSI), Tampa Scale of Kinesiophobia (TSK) and Global Perceived Effect questionnaire (GPE).

ELIGIBILITY:
Inclusion Criteria:

* men and women, between 16 and 45 years of age, minimum one traumatic anterior shoulder dislocation diagnosed with TASI, eligible for stabilizing Bankart surgery

Exclusion Criteria:

* complex shoulder injuries not suitable for a Bankart procedure as determined by an orthopedic surgeon, insufficient Norwegian language skills, and/or not being able to participate in a supervised exercise program

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Ontario Shoulder Instability Index (WOSI) | Baseline, 12 weeks
  change in shoulder quality of life

SECONDARY OUTCOMES:
Tampa Scale of Kinesiophobia (TSK) | Baseline, 12 weeks
  Change in fear of movement and re-injury, numbers
Sensorimotor control measured by center of pressure path length (COPL) | Baseline, 12 weeks
  Change in shoulder stability, mm
Shoulder joint position sense (SJPS) | Baseline, 12 weeks
  Change in shoulder position stability, degrees
Isometric strength measured by Constant Score - Isometric Maximal Voluntary Contraction (CS-iMVC) | Baseline, 12 weeks
  Change in muscle strength, kg
Apprehension and relocation tests | Baseline, 12 weeks
  Change in anterior glenohumeral instability, positive/negative
Global Perceived Effect questionnaire (GPE) | at 12 weeks
  Impression of change, 1-7

CONTACTS AND LOCATIONS:
Overall Officials: Gro Anita F Flaten, ph.d., Study Director — Western Norway University of Applied Sciences
Locations (1):
- Bergen University College, Bergen, Norway

REFERENCES:
- [Derived] Hagesaeter AN, Lovold T, Juul-Kristensen B, Blomquist J, Hole R, Eshoj H, Magnussen LH. Feasibility of the SINEX program for patients with traumatic anterior shoulder instability. Pilot Feasibility Stud. 2020 Oct 6;6:148. doi: 10.1186/s40814-020-00679-x. eCollection 2020. PMID 33042568